CLINICAL TRIAL: NCT03257020
Title: The Comparison of Bruch's Membrane Opening-minimum Rim Width and Retinal Nerve Fiber Layer Thickness and Their Combinational Index Using Artificial Neural Network
Brief Title: The Diagnostic Performance of BMO-MRW and RNFL Thickness and Their Combinational Index Using Artificial Neural Network
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1510-001-034
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma; Tomography, Optical Coherence
Keywords: OCT; RNFL; BMO-MRW; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal subject: Measure BMO-MRW and RNFL with SD-OCT. If the BMO-MRW and RNFL is within the normal range and those with no history of ocular disease, an intraocular pressure < 21 mmHg, an absence of glaucomatous optic disc appearance, and a normal visual field, they will be classified into normal group.
  Interventions: Diagnostic Test: SD-OCT
- Glaucoma patients: Measure BMO-MRW and RNFL with SD-OCT. If the BMO-MRW and RNFL is below the normal range and those with glaucomatous optic disc and two consecutive abnormal visual field test results with open angles on gonioscopy, glaucomatous optic neuropathy, RNFL defects congruent with visual field defects, they will be classified into glaucoma patients.
  Interventions: Diagnostic Test: SD-OCT

INTERVENTIONS:
Diagnostic Test: SD-OCT — SD-OCT was performed to all subjects to measure BMO-MRW and RNFL thickness by trained glaucoma specialist. It takes about 5 to 10 minutes. The foveal location was manually detected with a live B-scan, followed by defining BMO center. A radial pattern containing 24 angular, equidistant, high-resolution 15° B-scans centered on the BMO was used to compute the neuroretinal rim parameters. The BMO points and ILM were identified and marked in each B-scan with automated software (Glaucoma Module Premium Edition, version 6.0; Heidelberg Engineering). After radial scan completed, 3 consecutive circumpapillary B-scans were followed to measure RNFL thickness at diameter of 3.5, 4.1 and 4.7mm. BMO-MRW and RNFL thickness was automatically computed globally and sectorally.

SUMMARY:
This study evaluates the relationship between BMO-MRW and RNFL thickness measured by OCT. SD-OCT exam will be performed to all patients in this study.

DETAILED DESCRIPTION:
spectral domain optical coherence tomography, SD-OCT, (Heidelberg Engineering, Heidelberg, Germany) is a widely used commercial device in ophthalmology field. For a long time, retinal nerve fiber layer (RNFL) thickness was measured with OCT to detect and follow up glaucoma patients. Bruch's membrane opening - minimum rim width (BMO-MRW) is relatively new parameter which measures the minimum distance between Bruch's membrane opening to internal limiting membrane (ILM). BMO-MRW,a new parameter, is known to have better diagnostic performance than RNFL thickness and recently, many researches has been performed on this new parameter. SD-OCT can measure RNFL thickness and BMO-MRW at the same time. The test procedure is not different from RNFL thickness measurement but only software implemented in OCT device calculates BMO-MRW as well as RNFL thickness. The investigators are going to compare these two parameters and find out the relationship between two parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years with a clear cornea and clear ocular media
* BCVA ≥ 20/40
* Refractive error within ± 6.0 diopters (D) of 0 and astigmatism ± 3.0 D of 0

Exclusion Criteria:

* uveitis
* secondary glaucoma
* corneal abnormalities
* non-glaucomatous optic neuropathies
* previous trauma
* ocular surgery or laser treatment
* any other eye disease except glaucoma.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients who visited Pusan National University Hospital glaucoma clinic.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Bruch's membrane opening - minimum rim width (BMO-MRW) | 5~10 minutes
  SD-OCT will be performed to the patients to measure BMO-MRW by trained glaucoma specialist.

SECONDARY OUTCOMES:
Retinal nerve fiber layer (RNFL) thickness | 5~10 minutes
  SD-OCT will be performed to the patients to measure RNFL thickness. This is measured at the same time as BMO-MRW, not separately.

CONTACTS AND LOCATIONS:
Overall Officials: Jiwoong Lee, M.D., Ph.D, Principal Investigator — Medical Research Institute, Pusan National University Hospital, Busan, Korea
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for all primary and secondary outcome measures will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within 12 months after study published.
Access Criteria: Data access requests will be reviewed by an external independent review panel (PNUH IRB) and if they approve, data will be provided.